CLINICAL TRIAL: NCT00254345
Title: Effect of Provisional-Crown Surface Coating on Biofilm Formation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 191056HMO-CTIL
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Dental Plaque
Keywords: biofilm; adhesion; liquid polish; bonding resin; PMMA Polymethylmetacrylate; provisional crown; no antibiotics treatment three months prior to experiment; no mouth rinse with oral solutions one month prior to experiment
MeSH Terms: conditions — Dental Plaque; Tissue Adhesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: coating a dental restoration material ,polymethylmethacrylate, with liquid polish resin

SUMMARY:
Auto polymerizing poly methyl methacrylate (PMMA), and light initiated resin modified PMMAs, are commonly used for fabricating provisional restorations (PRs) during prosthetic treatment 1. Biofilm accumulated on these PRs may cause caries and inflammation of the surrounding tissue, tempering the outcome of the final restoration 2. Plaque adherence to temporary restorations was significantly increased compared with the untreated reference teeth 3. Biologic and physical properties of the various materials used as PRs were studied extensively 4-8 whereas their interaction with bacterial biofilm in vivo and ex vivo is less characterized.

One improvement in provisional restorative materials is the use of liquid polish. It is claimed that these materials gives a high luster finish to provisional bis-acryl restorations and processed acrylic appliances, reduces or eliminates costly and time consuming polishing steps and can be used on all types of direct and indirect restorations and appliances.The effect of liquid polish coating or resin bonding coating on biofilm formation on PRs was not reported.

DETAILED DESCRIPTION:
Auto polymerizing poly methyl methacrylate (PMMA), and light initiated resin modified PMMAs, are commonly used for fabricating provisional restorations (PRs) during prosthetic treatment 1. Biofilm accumulated on these PRs may cause caries and inflammation of the surrounding tissue, tempering the outcome of the final restoration 2. Plaque adherence to temporary restorations was significantly increased compared with the untreated reference teeth 3. Biologic and physical properties of the various materials used as PRs were studied extensively 4-8 whereas their interaction with bacterial biofilm in vivo and ex vivo is less characterized.

One improvement in provisional restorative materials is the use of liquid polish. It is claimed that these materials gives a high luster finish to provisional bis-acryl restorations and processed acrylic appliances, reduces or eliminates costly and time consuming polishing steps and can be used on all types of direct and indirect restorations and appliances.

The effect of liquid polish coating or resin bonding coating on biofilm formation on PRs was not reported. In this study we intend to measure, in vivo early biofilm formation on PMMA PRs with and without resin coatings.

ELIGIBILITY:
Inclusion Criteria:

* Patient in need for PMAA provisional crowns

Exclusion Criteria:

* Patient took antibiotics three months prior to experiment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1
Dates: Start 2006-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
surface coating with reduced biofilm formation demonstrated by confocal scanning laser microscope and scanning electron microscope

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Perez Davidi, DMD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel

REFERENCES:
- [Result] Perez Davidi M, Beyth N, Sterer N, Feuerstein O, Weiss EI. Effect of liquid-polish coating on in vivo biofilm accumulation on provisional restorations: part 1. Quintessence Int. 2007 Jul-Aug;38(7):591-6. PMID 17694216
- See also: Michael Perez Davidi — http://www.mypd.co.il